CLINICAL TRIAL: NCT06367491
Title: Banca Dati Nazionale Metastasi Ossee
Brief Title: National Database of Bone Metastases
Acronym: BDMO
Status: Recruiting | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST100.12
Record Dates: First submitted 2024-03-13; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Bone Metastases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with bone metastasis: All patients with bone metastasis
  Interventions: Other: Registration in a database

INTERVENTIONS:
Other: Registration in a database — All patients with bone metastasis enrolled at the centre will be entered into the database and followed until death or interruption of follow-up for any another cause

SUMMARY:
BDMO is an Italian multicentre, observational, prospective study that collects data from all patients with bone metastases referred to each participating centre, using an on-line software 'tailor-made' for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Radiological and/or histological diagnosis of bone metastasis from histologically established solid tumor
* Males or females aged >= 18 years
* Informed consent

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bone metasis in any site.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-10-08 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
The establishment of a National Bone Metastasis Database at the IRCCS IRST | Up to 15 years

SECONDARY OUTCOMES:
Evaluation of clinical factors related to the primary tumor and metastases | Up to 15 years
  Descriptive statistics will be calculated on the basis of the stratification factors identified at baseline assessment (age, sex, site and morphology of primary tumour, number of lesions, type of metastasis)
Evaluation of clinical factors related to the primary tumor and metastases | Up to 15 years
  Overall survival will be calculated as the time between the date of diagnosis of the primary tumour and death or the end of follow-up
Evaluation of clinical factors related to the primary tumor and metastases | Up to 15 years
  Disease-free interval will be calculated from the date of diagnosis of the primary tumour until the diagnosis of bone metastasis
Impact of treatment on skeletal events (SRE) | Up to 15 years
  Time to first skeletal related events (SRE) will be calculated from the date of incidence of the bone metastasis to the date of incidence of the first SRE, regardless of the type
Analysis of overall efficiency of the mono- and multidisciplinary pathway on skeletal events (SRE) | Up to 15 years
  The Skeletal Morbidity Rate (SMR) will be calculated by summing the SREs occurring during the observation period, for each patient
Evaluation of biological factors related to the primary tumour and metastases | Up to 15 years
  Evaluation of site-specific receptors

CONTACTS AND LOCATIONS:
Locations (30):
- Italy (30):
  - A.U.S.L. Imola, Imola, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - Osp. "Sacro Cuore di Gesù", Gallipoli, Lecce
  - Osp. S. Vincenzo - ASP Messina, Taormina, Messina
  - Osp. Ramazzini di Carpi - AUSL Modena, Carpi, Modena
  - P.O. "S. Maria delle Grazie", Pozzuoli, Napoli
  - Osp. degli Infermi, Faenza, Ravenna
  - Ospedale Umberto I, Lugo, Ravenna
  - Istituto Neurotraumatologico Italiano (INI), Grottaferrata, Roma
  - A.O.U. Ospedali Riuniti, Ancona
  - Centro di Riferimento Oncologico - IRCCS CRO, Aviano
  - A.O.U.C. Policlinico di Bari Osp."Giovanni XXIII", Bari
  - A.O. "S. Pio", Benevento
  - IRCCS Ist. Ortopedico Rizzoli, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - A.O. S. Croce e Carle, Cuneo
  - A.O.U. "Arcispedale S. Anna" - AUSL Ferrara, Ferrara
  - Ospedale Civile di Legnano - ASST Ovest Milanese, Legnano
  - Fond. IRCCS Istituto Nazionale dei Tumori - INT, Milan
  - A.O.R.N. "A. Cardarelli", Napoli
  - Istituto Oncologico Veneto, Padua
  - Fond. IRCCS Policlinico San Matteo, Pavia
  - Osp. Guglielmo da Saliceto, Piacenza
  - Osp. S. Maria delle Croci, Ravenna
  - IRCCS Arcispedale S. Maria Nuova - A.O. Reggio Emilia, Reggio Emilia
  - Ospedale degli Infermi, Rimini
  - IRCCS Fond. Policlinico "A. Gemelli" - U.O.C. Oncologia Medica, Roma
  - IRCCS Fond. Policlinico "A. Gemelli" - U.O.S. Senologia Medica / U.O.C. Ginecologia oncologica, Roma
  - Ospedale di Treviglio - Caravaggio ASST Bergamo Ovest, Treviglio
  - A.O.U.I. Verona, Verona

IPD SHARING:
Plan to Share IPD: No